CLINICAL TRIAL: NCT06681311
Title: The Effects of Core and Shoulder Stabilization Exercises on Athletic Performance and Injury Risk in Master Swimmers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MarmaraU- AYDOĞDU- ÇETİN001
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-07

CONDITIONS: Athletic Performance and Injury Risk
Keywords: Master Swimmers; Stabilization Exercises; Athletic Performance; Injury Risk Assesment
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercises Group (Experimental)
  Interventions: Other: Exercises
- Control Group (No Intervention)

INTERVENTIONS:
Other: Exercises — During the research period, all participants will undergo swimming training for 1 hour per day, 3-4 days a week for 6 weeks. The control group will perform a 5-minute land warm-up covering traditional shoulder, torso, and leg areas before their routine swimming training. In addition to the traditional warm-up program and swimming training, the experimental group will also participate in core and shoulder stabilization exercises under the supervision of a physiotherapist.
  Arms: Exercises Group

SUMMARY:
The inclusion of dryland training and stabilization exercises is crucial for optimizing performance and reducing injury risk in master swimmers. Exercises targeting core stabilization play a significant role in enhancing overall body strength and endurance, thereby improving swimming performance. Shoulder stabilization exercises address common issues faced by swimmers, such as shoulder impingement and rotator cuff injuries, contributing to the prevention of such injuries. Incorporating these exercises into the training regimen enables master swimmers to improve their posture, balance, and strength, resulting in more efficient performance in the water and reduced injury risk. Thus, a comprehensive training approach that includes both aquatic and stabilization exercises is of great importance for sustaining performance and ensuring long-term health in master swimmers.

The aim of this study is to examine the effects of core and shoulder stabilization exercise training on athletic performance and injury risk in master swimmers. Our study is designed to include healthy swimmer participants. A minimum of 34 master swimmers aged between 25 and 50 years will be recruited for the study. Prior to the stabilization training program, participants will undergo several assessments including the Isometric Plank Test (Prone Bridge Test), Closed Kinetic Chain Test, Medicine Ball Throw Test, 50m Freestyle Test, and Functional Movement Screening for injury risk assessment. After initial testing, the control group will perform a 5-minute traditional dryland warm-up focusing on the shoulders, core, and lower extremities before swimming workouts. The experimental group will receive core and shoulder stabilization exercises in addition to the traditional dryland warm-up and routine swimming training for 6 weeks (2 days per week). To assess the effects of the intervention, all tests will be repeated at the beginning, at the end of the 6-week exercise program, and in the 12th week. The literature does not provide information on the relationship between combined core and shoulder stabilization exercises and performance or injury risk in swimmers. This study aims to address this gap in the literature by investigating whether there are significant differences in the results obtained from the exercises and to contribute to future research aimed at enhancing performance and reducing injury risk in athletes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 25-50
* Those who engage in swimming training at least 3-4 days a week
* Volunteers willing to participate in the study
* Licensed competitive swimmers
* Masters swimmers (A competitive swimming class for swimmers aged 25 and older, knowledgeable in swimming techniques and competing according to FINA (International Swimming Federation) rules) (https://www.worldaquatics.com/masters/latest; Accessed: 25.05.2024)

Exclusion Criteria:

* Individuals with chronic diseases affecting orthopedic, neurological, cardiovascular, or other systems
* Individuals with cognitive dysfunction
* Those who regularly engage in strength training
* Non-volunteers unwilling to participate in the study
* Individuals outside the age range of 25-50
* Any condition or discomfort that would hinder the performance of tests
* Having sustained a sports injury affecting swimming performance in the past six months

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Functional Movement Screen | At the baseline
  The evaluation of injury risk in participants will be conducted purposefully. The Functional Movement Screening (FMS) will be used for this assessment (Lockie et al., 2015). The FMS consists of seven fundamental movements: deep squat, hurdle step, inline lunge, shoulder mobility, active straight-leg raise, trunk stability push-up, and rotary stability (Cook et al., 2006). Scoring will be performed based on observations: a score of 3 will be given when the movement is performed in the desired pattern, 2 points if the movement is partially or fully completed but with compensatory mechanisms used, 1 point if the movement is not completed, and 0 points if pain is present at any point during the movement. The total score for the athlete will be calculated by summing the scores obtained from each movement. If the athlete scores 14 or less, their functional movement capacity will be defined as low and the risk of injury will be considered high (Cook et al., 2006).
Functional Movement Screen | Six week later
  The evaluation of injury risk in participants will be conducted purposefully. The Functional Movement Screening (FMS) will be used for this assessment (Lockie et al., 2015). The FMS consists of seven fundamental movements: deep squat, hurdle step, inline lunge, shoulder mobility, active straight-leg raise, trunk stability push-up, and rotary stability (Cook et al., 2006). Scoring will be performed based on observations: a score of 3 will be given when the movement is performed in the desired pattern, 2 points if the movement is partially or fully completed but with compensatory mechanisms used, 1 point if the movement is not completed, and 0 points if pain is present at any point during the movement. The total score for the athlete will be calculated by summing the scores obtained from each movement. If the athlete scores 14 or less, their functional movement capacity will be defined as low and the risk of injury will be considered high (Cook et al., 2006).
Functional Movement Screen | Twelve week later
  The evaluation of injury risk in participants will be conducted purposefully. The Functional Movement Screening (FMS) will be used for this assessment (Lockie et al., 2015). The FMS consists of seven fundamental movements: deep squat, hurdle step, inline lunge, shoulder mobility, active straight-leg raise, trunk stability push-up, and rotary stability (Cook et al., 2006). Scoring will be performed based on observations: a score of 3 will be given when the movement is performed in the desired pattern, 2 points if the movement is partially or fully completed but with compensatory mechanisms used, 1 point if the movement is not completed, and 0 points if pain is present at any point during the movement. The total score for the athlete will be calculated by summing the scores obtained from each movement. If the athlete scores 14 or less, their functional movement capacity will be defined as low and the risk of injury will be considered high (Cook et al., 2006).

SECONDARY OUTCOMES:
Prone Bridge Test | At the baseline
  To assess participants' core endurance, an isometric plank test will be administered. Participants will be instructed to assume a push-up position with their elbows directly beneath their shoulders, forearms, and fingers extended straight ahead. The body should remain straight from the head to the heels, and the neck should be in a neutral position (Tong et al., 2014). When the participant reaches the correct position, the timer will start immediately. The test will be terminated if the participant cannot maintain a straight back or if the hips drop. The duration will be recorded in minutes and seconds using a stopwatch. The goal of this test is to hold the high position for as long as possible (Bohannon et al., 2018).
Prone Bridge Test | Six week later
  To assess participants' core endurance, an isometric plank test will be administered. Participants will be instructed to assume a push-up position with their elbows directly beneath their shoulders, forearms, and fingers extended straight ahead. The body should remain straight from the head to the heels, and the neck should be in a neutral position (Tong et al., 2014). When the participant reaches the correct position, the timer will start immediately. The test will be terminated if the participant cannot maintain a straight back or if the hips drop. The duration will be recorded in minutes and seconds using a stopwatch. The goal of this test is to hold the high position for as long as possible (Bohannon et al., 2018).
Prone Bridge Test | Twelve week later
  To assess participants' core endurance, an isometric plank test will be administered. Participants will be instructed to assume a push-up position with their elbows directly beneath their shoulders, forearms, and fingers extended straight ahead. The body should remain straight from the head to the heels, and the neck should be in a neutral position (Tong et al., 2014). When the participant reaches the correct position, the timer will start immediately. The test will be terminated if the participant cannot maintain a straight back or if the hips drop. The duration will be recorded in minutes and seconds using a stopwatch. The goal of this test is to hold the high position for as long as possible (Bohannon et al., 2018).
Closed Kinetic Chain Test | At the baseline
  The Closed Kinetic Chain (CKC) test will be administered to assess the upper extremity stability of participants. To perform the test, men will assume a push-up position, while women will take a modified push-up position (knee push-up). Both will place their hands on two strips of tape spaced 91.4 cm (36 inches) apart, with the third finger touching the ground (Tucci et al., 2017). Participants must keep their bodies as straight as possible while maintaining their weight on the upper extremities. To start the test, the participant moves one hand from the tape line to the other side, touches the other hand, and then returns to the original line. The process is then repeated with the other hand, and this is done as many times as possible in 15 seconds (Tucci et al., 2017). The test is repeated three times with 45-second rest intervals between each attempt. The score will be calculated based on the arithmetic mean of the touches (de Oliveira et al., 2017).
Closed Kinetic Chain Test | Six week later
  The Closed Kinetic Chain (CKC) test will be administered to assess the upper extremity stability of participants. To perform the test, men will assume a push-up position, while women will take a modified push-up position (knee push-up). Both will place their hands on two strips of tape spaced 91.4 cm (36 inches) apart, with the third finger touching the ground (Tucci et al., 2017). Participants must keep their bodies as straight as possible while maintaining their weight on the upper extremities. To start the test, the participant moves one hand from the tape line to the other side, touches the other hand, and then returns to the original line. The process is then repeated with the other hand, and this is done as many times as possible in 15 seconds (Tucci et al., 2017). The test is repeated three times with 45-second rest intervals between each attempt. The score will be calculated based on the arithmetic mean of the touches (de Oliveira et al., 2017).
Closed Kinetic Chain Test | Twelve week later
  The Closed Kinetic Chain (CKC) test will be administered to assess the upper extremity stability of participants. To perform the test, men will assume a push-up position, while women will take a modified push-up position (knee push-up). Both will place their hands on two strips of tape spaced 91.4 cm (36 inches) apart, with the third finger touching the ground (Tucci et al., 2017). Participants must keep their bodies as straight as possible while maintaining their weight on the upper extremities. To start the test, the participant moves one hand from the tape line to the other side, touches the other hand, and then returns to the original line. The process is then repeated with the other hand, and this is done as many times as possible in 15 seconds (Tucci et al., 2017). The test is repeated three times with 45-second rest intervals between each attempt. The score will be calculated based on the arithmetic mean of the touches (de Oliveira et al., 2017).
Medicine Ball Throw Test | At the baseline
  This test will be used to assess the open kinetic chain function and explosive power of the participants' upper extremities. For the test, the athlete will be positioned with their back, shoulders, and head touching the wall. A 3 kg medicine ball will be held with both hands and positioned to touch the chest wall. The athlete will be instructed to throw the medicine ball as far as possible in a straight line with a chest pass, without breaking contact with the wall (Shinkle et al., 2012). The athlete will be instructed not to "swing back" or "pump" the ball before initiating the throw in order to minimize momentum and muscle variation (Sharrock et al., 2011). The medicine ball throw will be performed twice, and the best distance will be used for evaluation. The point where the ball first touches the ground will be marked and measured in meters. A 1-minute rest will be provided between each throw (Shinkle et al., 2012).
Medicine Ball Throw Test | Six week later
  This test will be used to assess the open kinetic chain function and explosive power of the participants' upper extremities. For the test, the athlete will be positioned with their back, shoulders, and head touching the wall. A 3 kg medicine ball will be held with both hands and positioned to touch the chest wall. The athlete will be instructed to throw the medicine ball as far as possible in a straight line with a chest pass, without breaking contact with the wall (Shinkle et al., 2012). The athlete will be instructed not to "swing back" or "pump" the ball before initiating the throw in order to minimize momentum and muscle variation (Sharrock et al., 2011). The medicine ball throw will be performed twice, and the best distance will be used for evaluation. The point where the ball first touches the ground will be marked and measured in meters. A 1-minute rest will be provided between each throw (Shinkle et al., 2012).
Medicine Ball Throw Test | Twelve week later
  This test will be used to assess the open kinetic chain function and explosive power of the participants' upper extremities. For the test, the athlete will be positioned with their back, shoulders, and head touching the wall. A 3 kg medicine ball will be held with both hands and positioned to touch the chest wall. The athlete will be instructed to throw the medicine ball as far as possible in a straight line with a chest pass, without breaking contact with the wall (Shinkle et al., 2012). The athlete will be instructed not to "swing back" or "pump" the ball before initiating the throw in order to minimize momentum and muscle variation (Sharrock et al., 2011). The medicine ball throw will be performed twice, and the best distance will be used for evaluation. The point where the ball first touches the ground will be marked and measured in meters. A 1-minute rest will be provided between each throw (Shinkle et al., 2012).
50 m Freestyle Swimming Test | At the baseline
  The 50 m freestyle swimming test will be administered to evaluate the swimming performance of the participants. Measurements will be conducted in a 25 m lane in a closed swimming pool. Before the test, athletes will perform land-based warm-up exercises and complete their warm-up with 200 m freestyle, 200 m kick drills, and 4x25 m sprint swimming (Soydan, 2006). The 50 m freestyle swimming performance will be tested with the athlete starting from the pool edge, pushing off the wall with both legs from within the water, without using a starting block. The stopwatch will be stopped as soon as the athlete touches the lane's edge.
50 m Freestyle Swimming Test | Six week later
  The 50 m freestyle swimming test will be administered to evaluate the swimming performance of the participants. Measurements will be conducted in a 25 m lane in a closed swimming pool. Before the test, athletes will perform land-based warm-up exercises and complete their warm-up with 200 m freestyle, 200 m kick drills, and 4x25 m sprint swimming (Soydan, 2006). The 50 m freestyle swimming performance will be tested with the athlete starting from the pool edge, pushing off the wall with both legs from within the water, without using a starting block. The stopwatch will be stopped as soon as the athlete touches the lane's edge.
50 m Freestyle Swimming Test | Twelve week later
  The 50 m freestyle swimming test will be administered to evaluate the swimming performance of the participants. Measurements will be conducted in a 25 m lane in a closed swimming pool. Before the test, athletes will perform land-based warm-up exercises and complete their warm-up with 200 m freestyle, 200 m kick drills, and 4x25 m sprint swimming (Soydan, 2006). The 50 m freestyle swimming performance will be tested with the athlete starting from the pool edge, pushing off the wall with both legs from within the water, without using a starting block. The stopwatch will be stopped as soon as the athlete touches the lane's edge.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided